CLINICAL TRIAL: NCT00005613
Title: A Prospective, Comparative Trial of Allogeneic Versus Autologous Stem Cell Transplantation for High Risk Lymphoma
Brief Title: Peripheral Stem Cell Transplantation in Treating Patients With Non-Hodgkin's Lymphoma or Hodgkin's Disease
Acronym: CBV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11306; MCC-11306 (Other: Moffitt Cancer Center); IRB-4250 (Other: University of South Florida IRB); NCI-G00-1746 (Other: National Cancer Institute)
Record Dates: First submitted 2000-05-02; First posted 2004-06-25 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Etoposide; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Transplant (Experimental): autologous hematopoietic progenitor cell transplant
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Drug: BCNU
- Allogeneic Transplant (Experimental): allogeneic hematopoietic progenitor cell trasnplant
  Interventions: Drug: cyclophosphamide; Drug: etoposide; Drug: BCNU

INTERVENTIONS:
Drug: cyclophosphamide — Cyclophosphamide will be given at a dose of 1500 mg/m2/day IV over 1.0 hour on days -6, -5, -4, and -3.
Drug: etoposide — Etoposide will be given at a dose of 600 mg/m2/day over 3.0 hours on days -6, -5, and -4.
  Other Names: vp-16
Drug: BCNU — BCNU will be given at a dose of 150 mg/m2/day in 500 cc D5W over 3.0 hours on days -6, -5, and -4
  Other Names: Carmustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with allogeneic or autologous peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to compare the effectiveness of allogeneic stem cell transplantation with that of autologous peripheral stem cell transplantation in treating patients who have non-Hodgkin's lymphoma or Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the relapse rate, progression free survival, and overall survival in patients with high risk non-Hodgkin's lymphoma or Hodgkin's disease treated with allogeneic vs autologous stem cell transplantation. II. Compare the toxicities (short and long term) of these 2 regimens in these patients.

OUTLINE: Cytoreductive therapy: Patients receive 3 courses of salvage chemotherapy (e.g., dexamethasone, high dose cytarabine, and cisplatin (DHAP); etoposide, methylprednisolone, high dose cytarabine, and cisplatin (ESHAP); fludarabine, mitoxantrone, and dexamethasone (FND)). Harvest: Patients with an HLA identical sibling donor are assigned to the allogeneic peripheral blood stem cell (PBSC) transplantation group. Patients without an HLA identical sibling are assigned to the autologous PBSC transplantation group. Allogeneic OR autologous PBSC are harvested. Conditioning regimen: Patients receive high dose chemotherapy comprised of cyclophosphamide IV over 1 hour on days -6 to -3 and carmustine IV over 3 hours and etoposide IV over 3 hours on days -6 to -4. PBSC are infused on day 0. Patients are followed weekly for 3 months, then monthly for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-Hodgkin's lymphoma that has relapsed or failed to achieve complete remission after first line induction chemotherapy Intermediate or high grade (including mantle cell, but excluding lymphoblastic disease) No more than 1 prior salvage chemotherapy regimen, e.g.: Dexamethasone, high dose cytarabine, and cisplatin (DHAP) Etoposide, methylprednisolone, high dose cytarabine, and cisplatin (ESHAP) Low grade No more than 2 prior salvage chemotherapy regimens, e.g.: Fludarabine, mitoxantrone, and dexamethasone (FND) ESHAP DHAP OR Histologically proven stage III or IV Hodgkin's disease that has relapsed or failed to achieve remission after combination induction chemotherapy Prior primary radiotherapy allowed if relapse is high risk (e.g., recurrence in radiation field, B symptoms, liver/marrow involvement) No more than 2 prior salvage chemotherapy regimens Allogeneic stem cell transplantation group: Availability of 6 antigen (A, B, and DR loci) HLA matched sibling donor No active CNS disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 15 to 55 Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and SGPT no greater than 3 times normal PT and PTT normal Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: LVEF at least 45% by MUGA scan or echocardiogram No myocardial infarction within the past 6 months No arrhythmias unless medically controlled Pulmonary: FEV1 at least 50% predicted DLCO at least 50% predicted Other: No diabetes mellitus or thyroid disease unless medically controlled No active serious infection HIV negative Not pregnant or nursing Negative pregnancy test

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 1996-03; Primary Completion 2006-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
relapse rate | 5 years
  determine relapse rate after allogeneic versus autologous hematopoietic progenitor cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Goldstein, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- United States (2):
  - Florida Cancer Specialists, Fort Myers, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida